CLINICAL TRIAL: NCT06019936
Title: A Randomized,Double-blind, Placebo Controlled, Multicenter Study to Evaluate the Safety and Efficacy of MT2004 Capsule in Treatment of Cholestatic and Mixed Drug Induced Liver Injury (DILI)
Brief Title: A Randomized,Double-blind, Placebo Controlled, Multicenter Study to Evaluate the Safety and Efficacy of MT2004 Capsule in DILI Subjects
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xi'An Aolitai Pharmaceutical Technology Co Ltd (Industry)
Responsible Party: Sponsor
Organization: Shaanxi Micot Pharmaceutical Technology Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MT2004-II-C01; CTR20232066 (Other: Center For Drug Evaluation, NMPA)
Record Dates: First submitted 2023-08-25; First posted 2023-08-31 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Drug-Induced Liver Injury; Cholestatic Liver Injury; Mixed Liver Injury
Keywords: Drug-Induced Liver Injury
MeSH Terms: conditions — Chemical and Drug Induced Liver Injury

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The study will be double-blinded for MT2004/matching placebo. The subjects and the clinical personnel involved in the collection, monitoring, revision, or evaluation of AEs, or personnel who could have an impact on the outcome of the study will be blinded with respect to the subject's treatment assignment (MT2004 or placebo).Blinding will be maintained until at least the clinical phase of the study is completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MT2004 Capsule (Experimental): The MT2004 Capsule will be orally used twice daily after meal for 12 weeks.
  Interventions: Drug: MT2004 Capsule
- MT2004 Capsule Placebo (Placebo Comparator): The MT2004 Capsule Placebo will be orally used twice daily after meal for 12 weeks.
  Interventions: Drug: MT2004 Capsule Placebo

INTERVENTIONS:
Drug: MT2004 Capsule — The stratified randomization method will be used in this study. In treatment period, the participants will orally receive the MT2004 (BID) for 12 weeks with the dose level of 25mg. The adjustment of the dose level will base on the decesion of Independent Data Monitoring Board (IDMC). The highest dose will not exceed the 50mg BID.
  Other Names: MT2004
  Arms: MT2004 Capsule
Drug: MT2004 Capsule Placebo — The stratified randomization method will be used in this study. In treatment period, the participants will orally receive the MT2004 Capsule Placebo (BID) for 12 weeks with the dose level of 25mg. The adjustment of the dose level will base on the decesion of Independent Data Monitoring Board (IDMC). The highest dose will not exceed the 50mg BID.
  Arms: MT2004 Capsule Placebo

SUMMARY:
The goal of this randomized, double-blind, placebo controlled, Multicenter Phase II clinical trial is to initially evaluate the Safety and Efficacy of MT2004 Capsule in Cholestatic and Mixed drug induced liver injury (DILI) subjects.

The main questions it aims to answer are:

1. The Efficacy of MT2004 Capsule in Cholestatic and Mixed DILI subjects
2. The Safety and Pharmacokinetic characteristic of MT2004 Capsule in Cholestatic and Mixed DILI subjects
3. The mechanism of using MT2004 Capsule on Cholestatic and Mixed DILI subjects

DETAILED DESCRIPTION:
Xi'An Aolitai Pharmaceutical Technology Co Ltd is developing MT2004, a novel investigational synthetic small molecule farnesoid X receptor (FXR) agonist targeted to the liver. The MT2004 was designed as the prodrug and the metabolites MT2004-met1 of MT2004 will act to the FXR receptor to regulate a series of genes expression. It also plays an important role in the metabolism of bile acids, lipids and sugars.

The goal of this randomized, double-blind, placebo controlled, Multicenter Phase II clinical trial is to initially evaluate the Safety and Efficacy of MT2004 Capsule in Cholestatic and Mixed drug induced liver injury (DILI) subjects. The whole study will be divied to three stages including screening period (14 Days before the treatment), treatment period (the participants will be randomized to receive MT2004, or placebo orally (BID), for 12 weeks) and follow-up period. The study aims to recruit total of 80 subjects with Cholestatic and Mixed DILI, in which 12 of subjects will be firstly enrolled and allocated to the MT2004 group (Dose level: 25mg) as well as control group with the proportion of 2:1 by using the stratified randomization method. During the whole study, the adjustment of the subjects amount, the dose level as well as randomization proportion will based on the decesion of Independent Data Monitoring Board (IDMC). The highest dose will not exceed the 50mg BID.

The placebo will be used in this study, and the researchers will compare the placebo and test article to see the safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* 1. 18≤ age ≤ 75 years, male or female.

  2. When diagnosis of acute DILI, the liver biochemical threshold of patients must meet one of the following criteria: ：(1) ALT ≥5 ×ULN；(2) ALP ≥2× ULN；(3) ALT≥3× ULN and TBil ≥2×ULN.

  3. ALP ≥2× ULN, and conform to the clinical classification of cholestatic type or mixed type DILI in the Chinese Guidelines for the Diagnosis and Treatment of Drug-induced Liver Injury (2023 edition) (cholestatic type: R value ≤2; Mixed type: 2<R value <5).

  4. Excluded other common causes of acute liver injury, such as acute viral hepatitis A, B, C, E, autoimmune hepatitis, biliary tract disease, PBC, etc. (Exclusive diagnostic tests completed in our hospital or other hospitals after this suspected acute DILI event or within 2 months before screening were acceptable)

  5. RUCAM causality scale score ≥6 points; If the RUCAM score is between the 3-5 it is necessary to evaluate the causal relationship by three experts according to the evaluation criteria of expert opinions in the Chinese Guidelines for the Diagnosis and Treatment of Drug-induced Liver Injury (2023 edition), and at least two experts determine that the liver injury of the patients are "likely", "very likely" or "definitely" caused by drugs.

  6. The serious level of DILI is within level 1-2 based on the Chinese Guidelines for the Diagnosis and Treatment of Drug-induced Liver Injury (2023 edition).

  7. The duration of this liver injury is less than 6 months.

  8. The female with fertility must have had a negative pregnancy test results before being enrolled, or at least 1 year after pausimenia, or permanent sterilization ≥6 weeks（There should have a recording of hysterectomy, bilateral salpingo-oophorectomy）. The female and their male partners with the fertility potential agree to utilize the effective contraceptive methods（the following two methods can be selected: 1. any of the condom, diaphragm, Sponge or Cervical Cap with with Spermicide ）.

  9. Fully understand the study process of the clinical trial, and provide the signed ICF of joinning the clinical trial.

Exclusion Criteria:

* 1. Acute or chronic liver failure or liver decompensation

  2. The history of liver decompensation or portal hypertension history

  3. Moderate or above renal insufficiency, creatinine clearance (Ccr) < 60mL/min (according to the MDRD formula).

  4. Patients with serious diabetes and had poor control of blood sugar (HbA1c>10%)

  5. Serious sysmetic diseases of cardiovascular, respiratory, neurological, urinary, digestive, and for any reason which, in the opinion of the Investigator think the subject is not suitable for participating in the study.

  6. The predict survival period < 6 months.

  7. Utilization of Perursodeoxycholic acid within 14 days before the treatment.

  8. Utilization of S-adenosylmethionine within 1 days before the treatment.

  9. The patients must regularly utilize the known strong CYP3A4/3A5 inhibitors such as Clarithromycin, Itraconazole, ketoconazole, Ritonavir, rifampicin, phenytoin, carbamazepine within 1 week before the treatment or for the whole study period.

  10. Allergies or intolerances to study drug ingredients

  11. Patients are under the gestation, lactation, or patients have the pregnancy planning during the study period and 90 days after the end of the clinical trial

  12. Patients are not willing to ban the alcohol during the study period.

  13. Patients had joined the other clinical trials within 3 months before the administration.

  14. Other conditions that the investigator think the subject is not suitable for participating in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-08-10 (Actual); Primary Completion 2025-08-10 (Estimated); Study Completion 2025-10-10 (Estimated)

PRIMARY OUTCOMES:
Primary efficacy endpoint | On the week 4 after the administration
  The efficacy of MT2004 will be evaluated based on the decreasing rate on serum ALP compared to baseline.

SECONDARY OUTCOMES:
Secondary efficacy endpoint | On the week 2,8,12 after the administration and the week 4 follow-up period
  The efficacy of MT2004 will be evaluated based on the decreasing rate on ALP compared to baseline.
Secondary efficacy endpoint | On the week 2,4,8,12 after the administration and the week 4 follow-up period
  The efficacy of MT2004 will be evaluated based on the percentage of patients whose ALP decreased by more than 15% from baseline.
Secondary efficacy endpoint | On the week 2,4,8,12 after the administration and the week 4 follow-up period
  The efficacy of MT2004 will be evaluated based on the recovery rate of ALP.
Secondary efficacy endpoint | On the week 2,4,8,12 after the administration and the week 4 follow-up period
  The efficacy of MT2004 will be evaluated based on the decreasing rate on GGT compared to baseline.
Secondary efficacy endpoint | On the week 2,4,8,12 after the administration and the week 4 follow-up period
  The efficacy of MT2004 will be evaluated based on the recovery rate of GGT.
Secondary efficacy endpoint | On the week 2,4,8,12 after the administration and the week 4 follow-up period
  The efficacy of MT2004 will be evaluated based on the decreasing rate on ALT compared to baseline.
Secondary efficacy endpoint | On the week 2,4,8,12 after the administration and the week 4 follow-up period
  The efficacy of MT2004 will be evaluated based on the recovery rate of ALT.
Secondary efficacy endpoint | On the week 2,4,8,12 after the administration and the week 4 follow-up period
  The efficacy of MT2004 will be evaluated based on the decreasing rate on AST compared to baseline.
Secondary efficacy endpoint | On the week 2,4,8,12 after the administration and the week 4 follow-up period
  The efficacy of MT2004 will be evaluated based on the recovery rate of AST.
Secondary efficacy endpoint | On the week 2,4,8,12 after the administration and the week 4 follow-up period
  The efficacy of MT2004 will be evaluated based on the decreasing rate on TBIL compared to baseline.
Secondary efficacy endpoint | On the week 2,4,8,12 after the administration and the week 4 follow-up period
  The efficacy of MT2004 will be evaluated based on the decreasing rate on TBA compared to baseline.
Secondary efficacy endpoint | On the week 2,4,8,12 after the administration
  The efficacy of MT2004 will be evaluated based on the area of serum ALP decreasing rate-time curve.
Secondary efficacy endpoint | On the week 2,4,8,12 after the administration and the week 4 follow-up period
  The efficacy of MT2004 will be evaluated based on the percentage of patients developed to DILI level 3-4 after the administration.

OTHER OUTCOMES:
Safety endpoint | From the date of screening until the date of last follow-up visit or early termination and end of study, assessed up to 12 weeks.
  Adverse Events（AEs) will be recorded and evaluated for their seriousness, severity, and relationship to the study drug.

CONTACTS AND LOCATIONS:
Overall Officials: YiMin Mao, Master, Principal Investigator — RenJi Hospital
Locations (1):
- Shanghai Jiaotong University School of Medicine,Renji Hospital, Shanghai, Shanghai Municipality, China